CLINICAL TRIAL: NCT06993701
Title: The Effect of Vimala Massage Applied by Parents on Infantile Colic, Sleep and Development Levels of Infants
Brief Title: Vimala Massage Infantile Colic, Sleep and Development Levels
Acronym: VIMCOLSLEEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kilis 7 Aralik University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Elif Simay KOÇ, Lecturer, Kilis 7 Aralik University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ataturk University
Record Dates: First submitted 2025-04-09; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Massage Effect
Keywords: vimala massage; infantile colic; sleep; developmental levels
MeSH Terms: conditions — Colic

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: 3 group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- mother massage group (Experimental): In family health centers, the time and hour of the massage training will be determined with the mothers of infants diagnosed with IC. At this stage, the researcher will provide face-to-face, applied, one-to-one training on massage to the mothers of the babies in the mother group according to the constructivist learning model. Each training will be explained specifically for the mother and her baby. The infant massage will be demonstrated by the researcher on the model, and the mother will be asked to apply it to her baby at the same time.
  Interventions: Behavioral: Vimala Massage Training for Mothers
- father massage group (Experimental): Unlike the mother group, in this group, one-to-one training will be given to the fathers of the babies. Each training will be explained specifically for the father and his baby.
  Interventions: Behavioral: Vimala Massage Training for Fathers
- Control group (Placebo Comparator): In the control group, only one of the parents, mother or father, who fulfills the inclusion criteria will participate.
  Interventions: Other: Control Intervention

INTERVENTIONS:
Behavioral: Vimala Massage Training for Fathers — Fathers will receive Vimala massage training and apply it regularly to their babies at home.
  Arms: father massage group
Other: Control Intervention — babies in the control group will not receive any intervention
  Arms: Control group
Behavioral: Vimala Massage Training for Mothers — Mothers will receive Vimala massage training and apply it regularly to their babies at home.
  Arms: mother massage group

SUMMARY:
Objective: The effect of Vimala massage applied by parents on infantile colic, sleep and developmental levels of infants will be investigated.

Method: The data of the randomised controlled study is planned to be conducted in 3 Family Health Centres in Kilis province between 01 Jun 2025-01 January 2026. The population of the study will consist of infants diagnosed with IC who come to the FHC centre for diagnosis, treatment or follow-up between the specified dates and meet the inclusion criteria.

DETAILED DESCRIPTION:
The sample size was calculated using the G*Power 3.1.9.7 software, and the required sample size was determined to be 66. To account for potential data loss, the sample size was increased by 10% for each group. As a result, 24 infants were planned for each group (mother massage group, father massage group, and control group), totaling 72 participants. Data will be collected using the Introductory Information Form, Infant Follow-up Form, Infant Colic Scale, Expanded Short Infant Sleep Questionnaire, Parent-Infant Caregiving Touch Scale, and the Massage Practice Competence Evaluation Form.

All data will be collected face-to-face by the researcher, who holds an instructor certificate from the International Association of Infant Massage (IAIM). After the pre-test data are collected, participants will be assigned to the relevant groups. No intervention will be applied to the infants in the control group.

Parents in the mother massage group and father massage group will attend Vimala Massage training sessions once a week for five weeks at pre-scheduled times at Family Health Centers (FHCs). At the end of the fifth week, parents in all groups (mother, father, and control) will be asked to complete the post-test data collection forms.

This study is supported by Atatürk University (Project No: TDK-2025-15472).

ELIGIBILITY:
Inclusion Criteria:

* Infants born at term (38-42 weeks of gestation)
* Aged between 1 and 3 months
* Birth weight between 2500 and 4500 grams
* No health problems other than infantile colic
* Growth and development percentile consistent with current age
* Diagnosed with infantile colic according to Rome IV criteria
* Not yet started any treatment for infantile colic
* No presence of diarrhea or constipation
* Parents with at least primary school education
* Able to speak and write in Turkish
* Provided written and verbal informed consent
* Volunteered to participate in the study

Exclusion Criteria:

Exclusion Criteria:

* Infants and parents who do not meet the inclusion criteria
* Infants with acute or chronic medical conditions (e.g., congenital anomalies, metabolic disorders)
* Infants currently receiving any pharmacological or complementary treatment for infantile colic
* Parents with communication difficulties or cognitive impairments that hinder comprehension of study procedures
* Parents who have previously participated in a similar infant massage or infantile colic intervention study
* Parents who are unable or unwilling to complete follow-up assessments or study procedures

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-21 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Infantile Colic Scale | 9 month
  The Infantile Colic Scale consists of 19 items rated on a 6-point Likert scale, ranging from 1 to 6. It is designed to assess the severity of colic symptoms in infants. Higher average scores on the scale indicate more severe colic symptoms, whereas lower averages suggest symptom reduction. The items are grouped under five subdimensions: cow's milk/soy protein allergy or intolerance, immature digestive system, underdeveloped central nervous system, difficult infant temperament, and issues related to parent-infant interaction.
Brief Infant Sleep Questionnaire-Revised | 9 month
  The Brief Infant Sleep Questionnaire-Revised (BISQ-R) includes 33 items and assesses infant sleep patterns based on parental reports from the past two weeks. The scoring framework comprises three expert-defined, conceptually grounded subscales. These subscales evaluate three distinct but interrelated aspects of infant sleep: (1) infant sleep behaviors (Infant Sleep), (2) parental perceptions of their child's sleep (Parental Perception), and (3) ecologically based parental behaviors known to influence sleep quality (Parental Behavior), each adjusted according to the infant's age. The total score ranges from 0 to 100, with higher scores indicating better overall sleep quality, more positive parental perceptions, and supportive parental practices that promote healthy sleep in infants.
Parent-Infant Caregiving Touch Scale | 9 month
  The Parent-Infant Caregiving Touch Scale (PICTS) is a 12-item self-report instrument designed to assess the frequency of affectionate and intentional touch behaviors expressed by parents toward their infants. It includes items evaluating how often the mother strokes areas such as the infant's back, head, abdomen, arms, and legs, as well as how frequently she holds, cuddles, rocks, kisses, and physically interacts with the baby. Responses are recorded using a 5-point Likert scale ranging from 1 ("Never") to 5 ("Very Often"). Higher scores indicate more frequent engagement in positive tactile caregiving behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Türkan KADİROĞLU, Asst. Prof. Dr., Study Director — Ataturk University
Locations (1):
- Atatürk Üniversty, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTICLE IS INTENDED TO BE SHARED AFTER IT IS PUBLISHED